CLINICAL TRIAL: NCT03587961
Title: Personalized Theratyping Trial
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: George Solomon (Other)
Responsible Party: Sponsor-Investigator, George Solomon, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001867; IMPACT-Solomon (Other: UAB)
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; lumacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Symdeko (Experimental): Patients who have a mutation that responds to a CFTR corrector from in vitro study will be given Symdeko, depending on the in vitro response pattern
  Interventions: Drug: Symdeko
- Ivacaftor (Experimental): Patients who have mutation response to a potentiator of CFTR function will be given Ivacaftor monotherapy.. Patients with a mutation equivalent to wild type will be given Ivacaftor.
  Interventions: Drug: Symdeko
- Orkambi (Experimental): Patients who have a mutation that responds to a CFTR corrector from in vitro study will be given Orkambi, depending on the in vitro response pattern
  Interventions: Drug: Symdeko

INTERVENTIONS:
Drug: Symdeko — explore the use of off-label CFTR modulators that may affect CFTR function in patients with CFTR mutations that are not currently approved for these drugs.
  Other Names: Orkambi; Ivacaftor

SUMMARY:
The purpose of this study is to explore the use of off-label CFTR modulators that may affect CFTR function in patients with CFTR mutations that are not currently approved for these drugs.

DETAILED DESCRIPTION:
The purpose of this study is to explore the use of off-label CFTR modulators that may affect CFTR function in patients with CFTR mutations that are not currently approved for these drugs. Symdeko (Tezacaftor/Ivacaftor), Orkambi (Ivacaftor and Lumacaftor), correctors of CFTR misfolding and Kalydeco (Ivacaftor), a potentiator of abnormal CFTR gating, will be explored as a treatment for patients with other CF mutations than those currently approved. Patients who have a mutation that responds to a CFTR corrector from in vitro study will be given Symdeko, or Orkambi, depending on the in vitro response pattern. Patients who have mutation response to a potentiator of CFTR function will be given Ivacaftor monotherapy. Patients with a mutation equivalent to wild type will be given Ivacaftor. If the patient is 6-12 years old, we will only study Orkambi or ivacaftor as symdeko is not yet FDA approved in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF
* Age ≥6 y.o.
* CFTR mutation that may respond to approved correctors/potentiators in the opinion of the study investigators
* Informed Consent/Assent
* Stable CF pulmonary regimen

Exclusion Criteria:

* Exacerbation requiring antibiotic or steroids for >28 days before trial entry
* Ongoing participation in a CFTR modulator study
* Active smoking in the past 6 months
* History of solid organ transplant
* Any condition which precludes the use of CFTR modulators: e.g. advanced cirrhosis, End-stage Renal Disease (ESRD)
* Any condition that precludes the patient from participation in the opinion of the investigator
* Any meds that have significant drug-drug interactions or any other off label use of CFTR modulators

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
spirometry | 32 weeks
  change in lung function as measured via spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No